CLINICAL TRIAL: NCT07363811
Title: Large Granular Lymphocytes as a Prognostic Factor in Metastatic Non-small Cell Lung Cancer Treated With Nivolumab
Brief Title: Large Granular Lymphocytes in mNSCLC Treated With Nivolumab
Status: Recruiting | Type: Observational
Sponsor: Necmettin Erbakan University (Other)
Responsible Party: Principal Investigator, Mehmet Artac, Chief of Medical Oncology Clinic, Prof. Dr., Necmettin Erbakan University
Other Study IDs: 26105/2025/5927
Record Dates: First submitted 2026-01-15; First posted 2026-01-23 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Metastatic NSCLC - Non-Small Cell Lung Cancer
Keywords: Large granular lymphocyte; Nivolumab
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Biospecimen Retention: Samples Without DNA — Venous blood samples will be collected immediately before starting nivolumab treatment and at the third month, and peripheral blood smears will be performed. Two hematology specialists will provide the percentage (%) of LGL cells. The specialists will be blinded to patient information and will not be able to see each other's results. Subsequently, the average of the results provided by the two specialists for each patient will be calculated.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Large granular lymphocytes (LGLs), which constitute 10-15% of peripheral blood mononuclear cells, are large lymphocytes with a round nucleus, large cytoplasm, and azurophilic granules in the cytoplasm.

Most normal LGLs in peripheral blood are natural killer (NK) cells, but some are T lymphocytes. These cells cannot be measured by a standard complete blood count (CBC) test. These cells, which can be detected by peripheral smear, are expressed numerically and as a percentage relative to other cells. The aim of this study is to determine the relationship between the percentage of LGLs at baseline and at three months and the response and clinical parameters in participants with metastatic non-small cell lung cancer treated with nivolumab in second-line therapy.

DETAILED DESCRIPTION:
Non-small cell lung cancer ranks first worldwide in 2022 in terms of both incidence and mortality when both genders are considered . Historically, the 5-year survival rate for patients with advanced non-small cell lung cancer (NSCLC) receiving chemotherapy was 5%. Effective treatment options for patients without targetable molecular alterations, especially those who progressed after first-line chemotherapy, were limited until recently. Immunotherapy checkpoint inhibitors, with clinically meaningful survival benefits, long-term responses, and favorable safety profiles compared to chemotherapy, have become the standard of care for patients who progress during or after platinum-based chemotherapy. Immune checkpoint inhibitors are also effective as first-line therapy and are recommended as standard treatment for untreated advanced NSCLC patients, either in combination with chemotherapy or without chemotherapy.

Nivolumab, a fully human, monoclonal, anti-programmed death-1 (PD-1) antibody, is the first PD-1 inhibitor to demonstrate clinically meaningful efficacy in NSCLC. Nivolumab is approved for second-line treatment of advanced NSCLC in patients with advanced squamous (CheckMate 017; NCT01642004) and non-squamous (CheckMate 057; NCT01673867) NSCLC, following platinum-based chemotherapy, compared to docetaxel, showing improved overall survival and a favorable safety profile. Pembrolizumab is a humanized IgG4 monoclonal antibody against programmed cell death protein 1 (PD-1). Phase 1 KEYNOTE-0018 and phase 2/3 KEYNOTE-0109 studies demonstrated a correlation between increased expression of the PD-1 ligand PD-L1 in patients with advanced non-small cell lung cancer and the benefit achieved with pembrolizumab treatment. KEYNOTE-024 is a study comparing pembrolizumab monotherapy as first-line treatment with platinum-based chemotherapy in 305 patients with metastatic non-small cell lung cancer and a PD-L1 tumor proportion score (TPS) of 50% or higher. Both progression-free survival and overall survival were significantly longer in the pembrolizumab group compared to the standard chemotherapy group (median 10.3 months and 6.0 months vs. 30.0 months and 14.2 months).

Large granular lymphocytes (LGLs) are large lymphocytes with a round or kidney-shaped nucleus, a large cytoplasm, and azurophilic granules in the cytoplasm. They constitute 10-15% of peripheral blood mononuclear cells. Most normal LGLs in peripheral blood are natural killer (NK) cells, but some are T lymphocytes. These cells cannot be measured by a normal hemogram test. These cells, which can be detected by peripheral smear, are expressed both numerically and as a percentage relative to other cells. It has been shown that an absolute decrease in lymphocyte count reduces the response to immunotherapy. However, there are no studies in the literature showing the relationship between LGL and immunotherapy response.

In this prospectively planned study, the investigators aim to investigate the relationship between LGL (large granular lymphocyte) levels at the start of treatment and at 3 months in participants with non-small cell lung cancer treated with anti-PD-1 (programmed cell death-1) and survival and clinical parameters.

ELIGIBILITY:
Inclusion Criteria:

* Histological and staging diagnosis of metastatic non-small cell lung cancer
* ECOG performance score between 0 and 2
* No contraindications for nivolumab

Exclusion Criteria:

* Patients diagnosed with mNSCLC who received nivolumab as adjuvant or perioperative therapy
* Those with a second primary malignancy undergoing active treatment
* Those who have not signed the informed consent form
* Those with additional hematological malignancies such as leukemia, lymphoma, or myelodysplastic syndrome
* Those who have undergone palliative or curative radiotherapy within the last three months
* Those with active viral/bacterial infections before nivolumab treatment
* Patients who have used steroids in the last three months

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with metastatic non-small cell lung cancer who were followed up at the Medical Oncology Clinic of Necmettin Erbakan University Hospital and treated with nivolumab as second-line therapy.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
Objective response rate according to RECIST 1.1 Evaluation of target lesions | From enrollment to the end of treatment at 12 weeks
  Complete Response (CR):
  Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm.
  Partial Response (PR): At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum of diameters.
  Progressive Disease (PD): At least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this may include the baseline sum). The sum must also demonstrate an absolute increase of at least 5 mm.
  Stable Disease (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD.

SECONDARY OUTCOMES:
Progression-free survival | From July 2025 to July 2027
  It was defined as the time from the initiation of nivolumab treatment until disease progression or death, whichever occurred first. For patients without progression, PFS was calculated from the date of data entry onwards.
Overall survival | From July 2025 to July 2027
  It was defined as the time from the start of nivolumab treatment until death from any cause, or until the last follow-up date for patients still alive.

CONTACTS AND LOCATIONS:
Overall Officials: Mehmet Artaç, Study Director — Necmettin Erbakan University Faculty of Medicine, Department of Medical Oncology
Locations (1):
- Necmettin Erbakan University Faculty of Medicine, Department of Medical Oncology, Konya, Meram, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Conroy MR, O'Sullivan H, Collins DC, Bambury RM, Power D, Grossman S, O'Reilly S. Exploring the prognostic impact of absolute lymphocyte count in patients treated with immune-checkpoint inhibitors. BJC Rep. 2024 Apr 18;2(1):31. doi: 10.1038/s44276-024-00058-6. PMID 39516713
- [Result] Oshimi K. Clinical Features, Pathogenesis, and Treatment of Large Granular Lymphocyte Leukemias. Intern Med. 2017;56(14):1759-1769. doi: 10.2169/internalmedicine.56.8881. Epub 2017 Jul 15. PMID 28717070
- [Result] Mok TSK, Wu YL, Kudaba I, Kowalski DM, Cho BC, Turna HZ, Castro G Jr, Srimuninnimit V, Laktionov KK, Bondarenko I, Kubota K, Lubiniecki GM, Zhang J, Kush D, Lopes G; KEYNOTE-042 Investigators. Pembrolizumab versus chemotherapy for previously untreated, PD-L1-expressing, locally advanced or metastatic non-small-cell lung cancer (KEYNOTE-042): a randomised, open-label, controlled, phase 3 trial. Lancet. 2019 May 4;393(10183):1819-1830. doi: 10.1016/S0140-6736(18)32409-7. Epub 2019 Apr 4. PMID 30955977
- [Result] Borghaei H, Gettinger S, Vokes EE, Chow LQM, Burgio MA, de Castro Carpeno J, Pluzanski A, Arrieta O, Frontera OA, Chiari R, Butts C, Wojcik-Tomaszewska J, Coudert B, Garassino MC, Ready N, Felip E, Garcia MA, Waterhouse D, Domine M, Barlesi F, Antonia S, Wohlleber M, Gerber DE, Czyzewicz G, Spigel DR, Crino L, Eberhardt WEE, Li A, Marimuthu S, Brahmer J. Five-Year Outcomes From the Randomized, Phase III Trials CheckMate 017 and 057: Nivolumab Versus Docetaxel in Previously Treated Non-Small-Cell Lung Cancer. J Clin Oncol. 2021 Mar 1;39(7):723-733. doi: 10.1200/JCO.20.01605. Epub 2021 Jan 15. PMID 33449799
- [Result] Reck M, Rodriguez-Abreu D, Robinson AG, Hui R, Csoszi T, Fulop A, Gottfried M, Peled N, Tafreshi A, Cuffe S, O'Brien M, Rao S, Hotta K, Leiby MA, Lubiniecki GM, Shentu Y, Rangwala R, Brahmer JR; KEYNOTE-024 Investigators. Pembrolizumab versus Chemotherapy for PD-L1-Positive Non-Small-Cell Lung Cancer. N Engl J Med. 2016 Nov 10;375(19):1823-1833. doi: 10.1056/NEJMoa1606774. Epub 2016 Oct 8. PMID 27718847
- [Result] Assi HI, Kamphorst AO, Moukalled NM, Ramalingam SS. Immune checkpoint inhibitors in advanced non-small cell lung cancer. Cancer. 2018 Jan 15;124(2):248-261. doi: 10.1002/cncr.31105. Epub 2017 Dec 6. PMID 29211297
- [Result] Bray F, Laversanne M, Sung H, Ferlay J, Siegel RL, Soerjomataram I, Jemal A. Global cancer statistics 2022: GLOBOCAN estimates of incidence and mortality worldwide for 36 cancers in 185 countries. CA Cancer J Clin. 2024 May-Jun;74(3):229-263. doi: 10.3322/caac.21834. Epub 2024 Apr 4. PMID 38572751